CLINICAL TRIAL: NCT05690542
Title: Nanoparticles in Blood: Understanding and Controlling Protein Corona for Optimized Nanomedicine
Acronym: NANOBLORONA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DEMAISTRE CNRS 2022
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Coagulation Tests
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients from intensive care units: patients with hemostasis disorders (coagulation and/or platelets), antiplatelet and/or anticoagulant treatment
  Interventions: Other: blood tests
- controls: healthy people
  Interventions: Other: blood tests

INTERVENTIONS:
Other: blood tests — evaluate the possible impact of iron oxide nanoparticles (superparamagnetic iron oxide = SPIONs) (N=10) in the blood circulation;

SUMMARY:
The main objective is to study the effect of engineered nanoparticles SPIONs (superparamagnetic iron oxide) on hemostasis. Nanoparticles will be incubated in blood and platelet aggregation will be measured. In parallel, nanoparticles will also be incubated in blood and then plasma proteins adsorbed on them will be separated and analyzed. The proteins found on the nanoparticles will be linked to the platelet aggregation observed to help developing innovative protein functionalized nanoprobes for optimized nanomedicine.

ELIGIBILITY:
Inclusion Criteria:

* all people

Exclusion Criteria:

* patient under 18 years old, legal protection measure, pregnancy

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Leftover plasma sample from controls and patients hospitalized in CHU Dijon
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
impact of nanoparticles on coagulation tests ou platelet functions | at the baseline

SECONDARY OUTCOMES:
Difference of behaviour of the nanoparticles (N=10 preparations) on coagulation cascade and platelet functions | at the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU DIJON BOURGOGNE - laboratoire mixte, Dijon, France